CLINICAL TRIAL: NCT02093767
Title: Open-Label Trial of a Prebiotic Preparation Containing Inulin and Oligofructose (Synergy-1) for the Treatment of Mild to Moderate Acute Ulcerative Colitis
Brief Title: Oligofructose-enriched Inulin for the Treatment of Mild to Moderate Active Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Crohn's and Colitis Canada (Other); Beneo GmbH (Industry)
Responsible Party: Principal Investigator, Levinus Dieleman, Professor, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MOP81396
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Ulcerative Colitis
Keywords: prebiotics; Synergy1
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7.5g dose Synergy1 (Active Comparator): 7.5 g/day dose of Synergy1 (oligofructose enriched inulin 1:1) for 9 weeks. The daily dose is dispersed in two sachets of 3.75 g each which are consumed at breakfast and dinner
  Interventions: Dietary Supplement: Synergy1
- 15g Synergy1 (Active Comparator): 15 g/day dose of Synergy1 (oligofructose enriched inulin 1:1) for 9 weeks. The daily dose is dispersed in two sachets of 7.5 g each which are consumed at breakfast and dinner
  Interventions: Dietary Supplement: Synergy1

INTERVENTIONS:
Dietary Supplement: Synergy1 — The prebiotic preparation, Synergy-1, consists of 1:1 inulin and oligosaccharide. The chicory derived inulin has a degree of polymerization (DP) of 10 to 60 (average DP of 25). The oligofructose is produced by partial enzymatic hydrolysis of chicory derived inulin and has a DP ranging between 3 and 7 (average DP of 4).

SUMMARY:
Based on the efficacy of inulin and oligofructose in treating experimental colitis and emerging evidence suggesting probiotics are efficacious in maintaining and inducing remission in human ulcerative colitis (UC), the investigators intend to conduct an open label study using Synergy-1, a 1:1 oligosaccharide/ inulin mixture, in patients with mild to moderately active left-sided UC. The investigators hypothesize that oligofructose-enriched inulin (Synergy-1) can be used safely in the treatment of mild to moderate UC, and daily oral administration of Synergy-1 will result in the clinical improvement and/ or remission of disease. Subjects will be randomized to either a 7.5g or 15g dose of Synergy-1 in order to investigate what amount of the prebiotic is efficacious and tolerable in patients with active UC. The clinical activity of disease will be evaluated using endoscopy and symptom scores. The investigators will also study the effect Synergy-1 on mucosal histology, intestinal microbiota composition and function and markers of inflammation (e.g. fecal calprotectin, cytokines). The study will be for 9 weeks from baseline wherein all subjects will receive Synergy-1 treatment. Half the subjects will receive a dose of 7.5g and half will receive 15g daily.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD) of the colon which manifests as mucosal inflammation and ulceration. The disease affects various lengths of the colon. It cycles through periods of symptomatic relapse and asymptomatic remission. During relapse, patients suffer from frequent passage of watery diarrhea which may contain blood and mucous. Currently pharmacological treatments of mild to moderate UC consist of 5 amino salicylic acid (5 ASA), corticosteroids, and immunosuppressive agents such as azathioprine (Imuran), its metabolite 6-mercaptopurine (6-MP) and cyclosporine. Although 5-ASA medications are well-tolerated and relatively safe, systematic reviews have shown that they are successful in inducing remission in 50% of patients. Systemic corticosteroids and immunosuppressive such as cyclosporine, azathioprine and 6-MP have considerable toxicity which can limit their use in some patients. Therefore alternatives to the current standard therapy are in search.

The pathogenesis of UC is thought to be due to a combination of genetic, environmental and immunological factors. Several studies have shown that among the environmental factors, commensal intestinal bacteria play an important role in the etiology of UC. Patients with UC demonstrate a general increase in bacterial mucosal adherence and inter-epithelial cell penetration. Mucosal biopsies from UC showed increased concentrations of potentially pathogenic strains of enterobacteria (Escherichia coli group), Bacteroides and Clostridium species, and a relative decrease in protective organisms such as Faecalibacterium and Bifidobacteria, as compared to healthy individuals.

In the search for treatments of UC that have a direct influence on bacterial factors, efforts have been directed at altering the composition of the intestinal microflora to favour more protective organisms such as Lactobacilli and Bifidobacteria, also called probiotic bacteria. Several probiotic formulas (VSL#3 and Mutaflor - E. coli Nissle 1917) have shown efficacy as induction or maintenance therapy for UC or pouchitis.

As an alternative to oral supplementation with probiotic bacteria, prebiotics are more easily produced and cost-effective substitute. Prebiotics are oligosaccharides that cannot be enzymatically hydrolyzed in the small intestine, however serve as substrates for fermentation by probiotic bacteria in the colon. Prebiotics occur in nature; inulin is derived from chicory and oligosaccharides are present in edible plants. Human studies with healthy volunteers consuming diet supplemented with oligofructose or inulin demonstrated significant increase in luminal bifidobacteria and the strict anaerobe Faecalibacterium prausnitzii. These colonic bacterial groups are shown to alter cytokine production toward a more anti-inflammatory profile such as stimulating dendritic cell IL-10 production. In addition fructo-oligosaccharides fermentation in the colon results in improved short-chain fatty acids (SCFA) production, and in particular butyrate, which is important for the energy metabolism, cell differentiation and regulation of the immune response in the colon. Ulcerative colitis (UC), a subset of Inflammatory Bowel Disease (IBD) is characterized by disturbed microbial community (dysbiosis) with marked decrease of strict anaerobes, in particular Faecalibacterium spp. and Roseburia ssp. in addition to lower production of SCFA. Based on these findings oligofructose-enriched inulin (Beneo™ Synergy1) was chosen to be used in this trial.

Primary Hypothesis: Synergy-1 is a prebiotic food ingredient that can be used safely in the treatment of mild to moderate UC, and daily oral administration of Synergy-1 will result in the clinical improvement and/ or remission of disease.

Secondary Hypothesis: The improvement of clinical disease from the daily oral administration of Synergy-1 correlates with:

* a decrease in inflammatory markers in biopsies (IL-1β, TNF-α) and feces (calprotectin),
* a modulation of the mucosal and luminal intestinal microbiota towards more protective bacteria and a decrease in potential pathogenic bacteria.

Objectives: This pilot study will evaluate if the use of Synergy-1 is safe, efficacious and tolerable for the treatment of active mild to moderate left-sided UC.

Treatment Endpoints:

1. Primary Endpoint: Clinical improvement defined as a decrease in the Mayo score of ≥ 3 but the total Mayo score remains ≥ 3.
2. Secondary Endpoint: Remission after 9 weeks of treatment (clinical and endoscopic remission is defined as a score of 0 in the rectal bleeding and stool frequency parts of the Mayo together with a score of 0 or 1 in the sigmoidoscopic portion of the Mayo. The total Mayo score must not be greater than 2.
3. Safety and Tolerability Endpoints:

   1. Tolerability: Withdrawal rate due to intolerable drug side effects including, but not limited to: unacceptable flatulence, abdominal rumbling, bloating, abdominal pain or diarrhea.
   2. Safety: Number of patients experiencing a toxic or severe adverse event (AE) during the treatment period as well as stool culture testing positive for intestinal pathogens.

Studies to Evaluate Mechanisms of Action of Synergy-1:

* Intestinal microflora changes in mucosal biopsies and fecal samples, using DGGE and 16S rDNA-tags pyrosequencing.
* Decrease in pro-inflammatory cytokines IL-1β and TNF- α mRNA, by RT PCR assay of colonic biopsies. Decrease of the amounts of calprotectin in feces.
* Short-chain fatty acids (SCFA) production and metabolism using gas chromatography (GC) and qRT-PCR for measurement of SCFA in stool, bacterial butyryl-CoA-transferase and monocarboxylate transporter 1 (MCT1) in mucosal samples.

Study Population: 25 individuals will be enrolled in this study. Subjects will be selected based on Inclusion and Exclusion criteria (see Eligible Criteria Session).

All patients who qualify and provide written consent will be randomized to receive 7.5g or 15g of Synergy-1.

Non-blinded Participation: As this is an open label study, the Investigator and the patients will know which group they are in.

Conduct of Subject Visits: All the information obtained during subject visits shall be reported in the subject's Source Document (SD).

"1." Screening Visit

* Obtainment of Informed Consent
* Medical History
* Hematology and Chemistry
* Stool Pathogens
* Pregnancy Test

"2." Baseline Visit Week 0

* Focused Physical Exam and Medical History
* Sigmoidoscopy
* Mayo Score Calculation
* Biopsies for Histology, Colonic Cytokine and Microflora analysis
* Fecal samples for Calprotectin and luminal microflora analysis
* Dispense Synergy-1
* Dispense Patient Diaries

"3." Visit at Treatment Week 3 and Week 6

* Telephone visit for Adverse Event and Compliance Monitoring
* Telephone visit for monitoring of filling-in the Patient Diaries
* Ask about food intake
* Ask about UC symptoms

"4." Visit at Treatment Week 9

* Focused Physical Exam
* Hematology and Chemistry
* Stool Pathogens
* Adverse Event Monitoring
* Sigmoidoscopy
* Ulcerative Colitis Disease Activity Index Calculation
* Biopsies for Histology, Colonic Cytokine and Microflora analysis
* Fecal samples for Calprotectin and luminal microflora analysis
* Compliance Monitoring
* Collection of the Patient Diaries
* Ask about food intake

Study Procedures: The following procedures will be conducted with results recorded in the Source Document (SD).

Safety Assessment and Consent

1. Obtainment of Informed Consent: Subjects will receive an information document about the study including the contact number of the principal investigator from the research nurse. After subjects have received the full information about expected benefits and possible side effects and inconveniences related to study participation, written consent will be obtained. The study will be explained by study investigators, and by the research nurse. The obtainment of informed consent will be documented in SD. Subject must commence study drug within 14 days of signing consent. Therefore, the screening visit and the Week 0 visit must be scheduled within 14 days so that eligible patients can be randomized and begin taking study drug.
2. Medical History: This will include evaluation of past and/or present conditions/surgical procedures associated with the following systems: cardiovascular, respiratory, gastrointestinal, renal, hepatic, endocrine/metabolic, neurologic, lymphatic, haematological, immune, musculoskeletal/ connective tissue, dermatological, genito-urinary, psychiatric function, or any other significant diseases or disorders. The research nurse will record all current concomitant medications as well as the UC treatments used by the patients in the last 6 months.
3. Physical Exam: Abbreviated physical examination will be performed by a physician at baseline and will include an examination of the following: general appearance, head, ears, eyes, nose, throat, neck and thyroid, skin, cardiovascular system, respiratory system, gastro-intestinal system, neurological system, musculoskeletal system and lymph nodes. Blood pressure and pulse rate will be obtained after the subject has remained in a sitting position for at least 3 minutes.
4. Focused Physical Exam: A focused examination of subject's abdomen will be conducted by palpating for tenderness and masses.
5. Hematology and Chemistry: Blood will be drawn for hemoglobin, serum creatinine, AST, alkaline phosphatase, bilirubin.
6. Stool Pathogens: A stool specimen will be taken to exclude enteric infection. Tests will include: Clostridium difficile toxin assay, ova and parasite and culture for Salmonella, Shigella, Campylobacter, and pathogenic E. coli 0157.
7. Serum Pregnancy Test: To exclude pregnancy, the research nurse will collect a blood sample at screening in women of childbearing age to test for β-HCG. The same sample used for chemistry may also be used for the pregnancy test.
8. Adverse Event Monitoring: Subjects will be questioned by the research nurse about any Severe Adverse Events.
9. Side Effect Monitoring: In the Side Effects section of the SD, the nurse will record the occurrence and severity of side effects: unacceptable flatulence, abdominal rumbling, bloating, abdominal pain or diarrhea thought to be related to the drug treatment.

Clinical Efficacy Assessment

1. Sigmoidoscopy: All sigmoidoscopies for one subject should be performed by the same investigator to eliminate inter-observer variability. After an enema preparation, subjects will undergo sigmoidoscopy. Mucosal appearance between the splenic flexure and the anal verge will be assessed, on a scale of 0 - 3. Pictures of the mucosa will be taken at this time. Retrospective results from a previous sigmoidoscopy or colonoscopy can be used in place of a baseline sigmoidoscopy provided the patient consents to be included in the study no later than 48h after the sigmoidoscopy/ colonoscopy has been done.
2. Calculating Mayo Score: Subject's symptoms for Mayo score calculation (rectal bleeding and stool frequency) will be assessed using verbal scoring based on subject recollection of symptoms. A score for each parameter will be calculated by taking the average of the scores for the last available 3 days prior to the study visit. Subjects will be questioned about symptoms both by the research nurse and the physician. The Mayo will be calculated by adding the individual scores of the four parameters - bowel frequency, rectal bleeding, endoscopic score and physician's rating of severity. If the score is 3 - 8 inclusive at week 0 and the inclusion/exclusion criteria were deemed appropriate at screening, the subject is eligible to initiate treatment.
3. Study Specimen Collection. Fecal samples and biopsies will be collected. Fecal samples will be assessed for fecal calprotectin and microbiota composition. This material will be snap frozen after collection. A total of 8 biopsies will be taken during sigmoidoscopy. For each type of analysis 2 biopsies will be taken from an area of disease between 15 and 20 cm from the anal verge. Biopsies will be used for analysis of mucosal host factors (qRT-PCR), mucosa-associated microbiota composition (16S pyrosequencing) and histology.
4. Compliance Monitoring at Study Visits: Subjects must bring in used and unused Synergy-1 sachets so they can be counted by the research nurse to assess compliance.

Dispensing of Study Materials

1. Dispensing of the Patient's Diaries: Each night the subject will record details of their UC symptoms from the previous 24 hours.
2. Dispensing of Synergy-1: The research nurse will verbally explain and provide a document directing how and when to take the Synergy1 supplementation. Subjects will be given a box by the research nurse with the amount of sachets required for 9 weeks of treatment.

Study Test Product, Dosages and Duration of Treatment

1. Investigational Product: The prebiotic preparation, Synergy-1, consists of 1:1 inulin and oligosaccharide. The chicory derived inulin has a degree of polymerization (DP) of 10 to 60 (average DP of 25). The oligofructose, which is produced by partial enzymatic hydrolysis of chicory derived inulin, is a mixture of β-fructans with a DP ranging between 3 and 7 (average DP of 4).
2. Dosage and Administration: Two doses of Synergy-1 will be tested, a low dose of 7.5 g/day and a high dose of 15 g/day. Synergy-1 will be supplied to subjects in sachets. It can be stored at room temperature. Subjects randomized to 15g per day will take 7.5g at breakfast only in week one. In week two, they will begin taking 7.5g at breakfast and 7.5g at dinner to reach the target dose of prebiotic. Subjects randomized to 7.5g per day will take a dose of 3.75g at breakfast only in week one. In week two they will begin taking 3.75g at breakfast and 3.75g at dinner throughout the study. The half dose in week one is intended to increase the tolerability of the compound. The powder will be mixed with a hot liquid to dissolve it and will be taken with meals.
3. Duration of Treatment: The duration of treatment will be 9 weeks.
4. Assessment of Compliance: The subject must return all used and unused Synergy-1 sachets so that they may be counted. Specific forms will be used to record treatment compliance in the Source Document. The subject must return their Patients Diaries.
5. Concomitant Treatments: Patients currently taking oral 5-ASA therapy will be continued on the drug at a stable dose. Dose must be stable for 2 weeks prior to the screening visit, and throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 65 years of age.
* Diagnosis of ulcerative colitis established by previous endoscopies, with histology and clinical course consistent with diagnosis.
* Colitis must extend for more than 15 cm above the anal verge, and involve at least the rectosigmoid.
* Mild to moderately active ulcerative colitis defined by a minimum score of 3 and a maximum score of 8 on the 12 point Mayo scale. Mayo scores are assigned by (1) stool frequency, (2) rectal bleeding, (3) endoscopic findings and (4) physician's overall assessment of disease severity
* At least one previous episode of ulcerative colitis, prior to the current episode
* Duration of current symptomatic episode less than 4 weeks.
* Ability to give valid informed consent.
* For females of childbearing potential, a negative pregnancy test.

Exclusion Criteria:

* Crohn's disease or pouchitis.
* Current infectious enteritis.
* Use of oral steroids within the last 4 weeks of the screening visit.
* Use of antibiotics within the last 2 weeks of the screening visit
* Change in dose of oral 5-ASA products within the last 2 weeks of the screening visit.
* Topical 5-ASA or steroids within 7 days prior to the baseline endoscopy
* Use of immunosuppressive or biological agent within 3 months of screening.
* Use of NSAIDS one week before screening.
* Use of anti-diarrheal drugs within the last 1 week of the screening visit.
* Use of probiotic preparations either prescribed or over-the-counter within two weeks of screening.
* Use of natural health products within 2 weeks of screening (except multivitamins and minerals)
* Significant hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease as determined by the investigator
* Imminent need for colectomy
* Presence of severe UC (defined as a Mayo of 9 or greater)
* Pregnancy or lactation
* Inability to give a valid informed consent or to properly comply with study procedures for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who show a decrease in the Mayo score ≥ 3 but the total Mayo score remains ≥ 3. | week 9
  Mayo score is a total of bowel frequency, rectal bleeding, endoscopic score and physician's rating of severity, each of the parameters on the scale 0-3.

SECONDARY OUTCOMES:
Number of patients who enter remission | week 9
  Clinical and endoscopic remission is defined as a score of 0 in the rectal bleeding and stool frequency parts of the Mayo together with a score of 0 or 1 in the sigmoidoscopic portion of the Mayo. The total Mayo score must not be greater than 2.

CONTACTS AND LOCATIONS:
Overall Officials: Levinus Dieleman, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No